CLINICAL TRIAL: NCT04867317
Title: CSP #2018 - Growth Hormone Replacement Therapy in Veterans With Mild Traumatic Brain Injury (mTBI) and Adult Growth Hormone Deficiency (AGHD)
Brief Title: Growth Hormone Replacement Therapy in Veterans With Mild Traumatic Brain Injury (mTBI) and Adult Growth Hormone Deficiency (AGHD)
Acronym: GRIT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018
Record Dates: First submitted 2021-04-08; First posted 2021-04-30 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Adult Growth Hormone Deficiency; Mild Traumatic Brain Injury
MeSH Terms: conditions — Dwarfism, Pituitary; Brain Concussion | interventions — Human Growth Hormone

STUDY DESIGN:
Intervention Model Description: Two arm study: active drug vs placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Growth Hormone Replacement Therapy (Active Comparator): Recombinant Human Growth Hormone
  Interventions: Drug: Somatropin
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Somatropin — Participants (n=172) will be randomized in a 1:1 ratio to rhGH (n=86) versus placebo (n=86) for six months, stratified by participating site. Both study participants and the study team will be blinded to treatment assignment. All participants will complete in-clinic follow-ups at Days 14, 40, 65, and 90 (3 months) and at day 180 (6 months). The primary outcome will be the mean difference in QoL-AGHDA scores between treatment arms at 6 months follow-up. Patients will discontinue the study intervention at 6 months, and will be followed-up two weeks subsequent, in order to assure patient safety and wellness, and to ensure maximal facilitation of patient transition back into routine care.
  Arms: Growth Hormone Replacement Therapy
Other: Placebo — Participants (n=172) will be randomized in a 1:1 ratio to rhGH (n=86) versus placebo (n=86) for six months, stratified by participating site. Both study participants and the study team will be blinded to treatment assignment. All participants will complete in-clinic follow-ups at Days 14, 40, 65, and 90 (3 months) and at day 180 (6 months). The primary outcome will be the mean difference in QoL-AGHDA scores between treatment arms at 6 months follow-up. Patients will discontinue the study intervention at 6 months, and will be followed-up two weeks subsequent, in order to assure patient safety and wellness, and to ensure maximal facilitation of patient transition back into routine care.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether growth hormone replacement therapy (GHRT) is effective versus placebo in the improvement of Quality of Life in patients with adult growth hormone deficiency (AGHD) and mild traumatic brain injury (mTBI).

ELIGIBILITY:
Inclusion Criteria:

* OEF/OIF/OND Veteran
* Score of 18 or more on Combat Experiences sub-scale of Deployment Risk and Resilience Inventory-2 (DRRI-2)
* Age 21 - 55 years old
* One or more mTBI sustained during military service at least 12 months prior to the screening date, as noted via the CRAFT survey
* GH deficiency diagnosed by: macimorelin stimulation test (cut point 5.1 mcg/L) and IGF-I lab values have to be less than or equal to +1 SDS at baseline
* Score of 11 or more on QoL-AGHDA
* 4-week stability on any psychotropic medications
* 3-month stability on all other hormone treatments
* Able and willing to provide informed consent to participate in this study, and complete study protocol.

Exclusion Criteria:

* History of moderate or severe TBI
* History of neurologic disorder other than TBI with substantial impact on quality of life
* History of bipolar disorder, schizophrenia, or other concurrent psychotic disorder
* Active suicidal ideation (no plan required) as determined by a score of 2 points or more on the Columbia Suicide Severity Rating Scale (C-SSRS) suicidal ideation rating, or overt suicidal behavior in the past 6 months
* Contraindication to rhGH therapy
* Contraindication to macimorelin use, including QTc interval >470ms
* Acute medical illness, active infection, cancer or decompensated chronic medical illness
* Evidence of substance use disorder, -other than mild alcohol or cannabis use disorder-, or urine toxicology evidence of the use of an illicit drug (excluding cannabis), in the past 6 months. Nicotine use is allowed.
* Score less than or equal to 41 on Trial 2 or Retention Trial of the Test of Memory Malingering (TOMM).
* BMI > 35 or body weight > 350 lbs
* Pituitary anatomy documented by an MRI using a sella protocol within the last 2 years indicating abnormalities consistent with an etiology other than mild-TBI (i.e.; pituitary mass)
* Women who are pregnant or of child-bearing potential not on contraception
* Current use of the following: growth hormone, estrogen or estrogen-like dietary supplements, progestin, IGF-I, or chronic glucocorticoid use in supraphysiologic doses
* Currently enrolled in any other interventional study unless prior approval is provided by the study chairs and the study sponsor (Cooperative Studies Program)

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 172 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
QoL-AGHDA (Quality of Life-Assessment of Adult Growth Hormone in Adults) | 6 months
  25 question survey on quality of life; The primary objective of CSP #2018 is to determine the efficacy of rhGH, given daily for 6 months, versus placebo to improve QoL, as measured by difference in mean QoL-AGHDA score, among Veterans with a history of mTBI and AGHD (primary outcome). The primary hypothesis is that the investigators, compared to placebo, patients treated with rhGH will exhibit a 3.5-point lower mean score (higher quality of life) in QoL-AGHDA at 6 months. QoL-AGHDA: minimum score=0 (high QoL: best outcome); maximum score=25 (low QoL: worst outcome).

SECONDARY OUTCOMES:
Body Composition | 6 months
  DEXA (Dual-Energy x-ray absorptiometry); The secondary objective of CSP #2018 is to investigate the efficacy of rhGH vs placebo on long-term surrogate outcomes: a) body composition, assessed through dual-energy x-ray absorptiometry (DEXA) and b) cardiometabolic risk factors including lipids, autonomic function, and highly sensitive C-reactive protein. The specific hypotheses for these outcomes are that compared to placebo there will be a 4.5% mean reduction in total truncal body fat percentage and a mean reduction of 10 mg/dL in LDL serum levels after 6 months of treatment and follow-up of rhGH.

OTHER OUTCOMES:
Depressive and Anxiety Symptoms measured by Depression Anxiety and Stress Scale (DASS-21) | 6 months
  Tertiary endpoint of interest: Depressive and anxiety symptoms measured by DASS-21 scores and post-traumatic stress symptoms measured by the PTSD Checklist for DSM-5 are expected to be lower (improved) within the rhGH arm after 6 months of therapy compared to the placebo arm.
Cognition | 6 months
  Tertiary endpoint of interest: Cognitive functioning will be assessed the Color Word Interference Test for cognitive flexibility and inhibition; the Digit Span test for working memory capacity; the Trail Making Test for processing speed, cognitive flexibility, and attention; the Grooved Pegboard for fine motor control and coordination; the Letter Fluency Test for verbal fluency and executive function; and the Rey Auditory Verbal Learning Test for verbal learning, memory, and attention. All test scores will be converted to z-scores, which standardize the results based on the mean and standard deviation of the normative sample, then averaged to generate a composite score, with higher scores indicating better performance relative to the normative sample. Both, individual test scores and the composite score will be analyzed to evaluate whether six-month recombinant human Growth Hormone treatment has any significant effect on cognitive performance.
Severity of Fatigue Symptoms | 6 months
  Tertiary endpoint of interest: Severity of fatigue symptoms measured by the Patient Health Questionnaire 15-item somatic symptom severity scale PHQ-15 are expected to improve after 6 months of rhGH therapy compared to the placebo arm.
Sleep Quality | 6 months
  Exploratory objective and hypothesis: Sleep quality as measured by the Pittsburgh Sleep Quality Index Score (PSQI). We hypothesize that subjective measures of sleep quality and daytime sleepiness will significantly improve in the active arm compared to placebo.
Chronic Pain Assessment | 6 months
  Exploratory objective and hypothesis: Chronic pain assessed using the Defense Veterans Pain Report System-II (DVPRS-II); hypothesize that pain severity and pain interference with activities of daily living will be significantly reduced among participants receiving GHRT compared to placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Jose M. Garcia, MD PhD, Study Chair — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (4):
- United States (4):
  - Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Digital data underlying primary scientific publications from this study will be held as part of a data sharing resource maintained by the Cooperative Studies Program (VA-CSP). These data may be available to the public and other VA and non-VA researchers under certain conditions and consistent with the informed consent and CSP policy which prioritize protecting subjects' privacy and confidentiality to the fullest extent possible.